CLINICAL TRIAL: NCT07256249
Title: Real-life Registry in Patients With Coronary Artery Disease Treated With the SELUTION Sirolimus-eluting Balloon. Selution Iberia Registry
Acronym: SELUTION
Status: Recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: rEPIC16- SELUTION
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Device: SELUTION SLRTM sirolimus coated balloon

INTERVENTIONS:
Device: SELUTION SLRTM sirolimus coated balloon — Patients in whom treatment with SELUTION SLRTM sirolimus coated balloon has been attempted

SUMMARY:
Selution Iberia registry is a post-market clinical follow-up, prospective, multicenter, international, longitudinal, observational study without a control group of consecutive unselected "real-world" patients with coronary artery disease in whom it was decided to use the SELUTION SLRTM device in the treatment of primary native lesions and ISR (in-stent restenosis) in all settings, in order to evaluate its effectiveness and safety.

The primary objective is to evaluate the effectiveness and safety of the Sirolimus-eluting balloon SELUTION SLRTM based strategy in the treatment of native coronary artery stenosis and in-stent restenosis. The primary endpoint will be the incidence of major adverse cardiovascular events at 12 months, including death, non-fatal myocardial infarction or target lesion revascularization for ischemia, in an unselected "real-world" patient setting. Both Device Oriented Composite Endpoint (Cardiovascular death, device failure-related myocardial infarction or device failure-related ischaemia) and Patient Oriented Composite Endpoint (all cause death, any stroke, any myocardial infarction or any revascularization) will be detailed.

DETAILED DESCRIPTION:
Selution Iberia registry is a post-market clinical follow-up, prospective, multicenter, international, longitudinal, observational study without a control group of consecutive unselected "real-world" patients with coronary artery disease in whom it was decided to use the SELUTION SLRTM device in the treatment of primary native lesions and ISR in all settings, in order to evaluate its effectiveness and safety.

The primary objective is to evaluate the effectiveness and safety of the Sirolimus-eluting balloon SELUTION SLRTM based strategy in the treatment of native coronary artery stenosis and in-stent restenosis. The primary endpoint will be the incidence of major adverse cardiovascular events at 12 months, including death, non-fatal myocardial infarction or target lesion revascularization for ischemia, in an unselected "real-world" patient setting. Both Device Oriented Composite Endpoint (Cardiovascular death, device failure-related myocardial infarction or device failure-related ischaemia) and Patient Oriented Composite Endpoint (all cause death, any stroke, any myocardial infarction or any revascularization) will be detailed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ≥18 years and;
* Patients with coronary artery disease in whom, at the operator's discretion, treatment of a lesion in a native vessel, coronary graft or coronary restenosis is decided using the Selution SLRTM device;
* Patient who has been informed of the characteristics of the study and has provided written informed consent.

Exclusion Criteria:

* Express refusal of the patient to participate in the study
* Life expectancy of the patient of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with the Selution SLRTM device
Sampling Method: Probability Sample
Enrollment: 960 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
MACE (Major Adverse Cardiovascular Events) | 12 months
  Incidence of MACE defined as death, nonfatal infarction, or need for TLR (Target Target Lesion Revascularization)
TLR | 12 months
  Number of Target Lesion Revascularizations
DoCE (Device-oriented Composite Endpoint) | 12 months
  Incidence of DoCE, defined as Cardiovascular death, device failure-related MI (Myocardial Infarction) or device failure-related ischaemia)
PoCE (Patient-oriented Composite Endpoint) | 12 months
  Incidence of PoCE defined as all cause death, any stroke, any MI or any revascularization

SECONDARY OUTCOMES:
TLR in ISR | 12 months
  Number of Target Lesion Revascularizations in patients with ISR (in-stent restenosis)
TLR in primary lesions in native vessel | 12 months
  Number of Target Lesion Revascularizations in primary lesions in native vessel
TLR in bifurcation side branch lesions | 12 months
  Number of Target Lesion Revascularizations in bifurcation side branch lesions
MACE (Major Adverse Cardiovascular Events) in ISR | 12 months
  Incidence of MACE defined as death, nonfatal infarction, or need for TLR (Target Target Lesion Revascularization) in ISR
MACE (Major Adverse Cardiovascular Events) in primary lesions in native vessel | 12 months
  Incidence of MACE defined as death, non fatal myocardial infarction, or need for TLR (Target Target Lesion Revascularization) in primary lesions in native vessel
MACE (Major Adverse Cardiovascular Events) in bifurcation side branch lesions | 12 months
  Incidence of MACE defined as death, nonfatal infarction, or need for TLR (Target Target Lesion Revascularization) in primary lesions in bifurcation side branch lesions
Procedure success | 1 day
  Device success defined as residual stenosis <30% by visual assessment and or online QCA (Quantitative Coronary Analysis) < 40%, absence of dissection and TIMI 3 flow
Death | 12 months
  Incidence of Death defined as all-cause, cardiac, device related, procedure related
Non fatal Myocardial Infarction | 12 months
  Incidence of Non fatal Myocardial Infarction

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitari MútuaTerrassa, Terrassa
  - Hospital Universitario de Torrevieja, Torrevieja

REFERENCES:
- [Background] Rittger H, Brachmann J, Sinha AM, Waliszewski M, Ohlow M, Brugger A, Thiele H, Birkemeyer R, Kurowski V, Breithardt OA, Schmidt M, Zimmermann S, Lonke S, von Cranach M, Nguyen TV, Daniel WG, Wohrle J. A randomized, multicenter, single-blinded trial comparing paclitaxel-coated balloon angioplasty with plain balloon angioplasty in drug-eluting stent restenosis: the PEPCAD-DES study. J Am Coll Cardiol. 2012 Apr 10;59(15):1377-82. doi: 10.1016/j.jacc.2012.01.015. Epub 2012 Feb 29. PMID 22386286
- [Background] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Leibundgut G, Weilenmann D, Wohrle J, Richter S, Schreiber M, Mahfoud F, Linke A, Stephan FP, Mueller C, Rickenbacher P, Coslovsky M, Gilgen N, Osswald S, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Drug-coated balloons for small coronary artery disease (BASKET-SMALL 2): an open-label randomised non-inferiority trial. Lancet. 2018 Sep 8;392(10150):849-856. doi: 10.1016/S0140-6736(18)31719-7. Epub 2018 Aug 28. PMID 30170854
- [Background] Costa RA, Mandal SC, Hazra PK, Chopda M, Chandra P, Damiani LP, Abizaid A, Hiremath S. Sirolimus-Coated Balloon With a Microsphere-Based Technology for the Treatment of De Novo or Restenotic Coronary Lesions. Cardiovasc Revasc Med. 2022 Dec;45:18-25. doi: 10.1016/j.carrev.2022.08.037. Epub 2022 Sep 5. PMID 36192319
- [Background] Madanchi M, Cioffi GM, Attinger-Toller A, Seiler T, Somm S, Koch T, Tersalvi G, Wolfrum M, Moccetti F, Toggweiler S, Kobza R, Levine MB, Garcia-Garcia HM, Bossard M, Cuculi F. Metal free percutaneous coronary interventions in all-comers: First experience with a novel sirolimus-coated balloon. Cardiol J. 2022;29(6):906-916. doi: 10.5603/CJ.a2022.0106. Epub 2022 Nov 17. PMID 36385601
- [Background] Spaulding C, Krackhardt F, Bogaerts K, Urban P, Meis S, Morice MC, Eccleshall S. Comparing a strategy of sirolimus-eluting balloon treatment to drug-eluting stent implantation in de novo coronary lesions in all-comers: Design and rationale of the SELUTION DeNovo Trial. Am Heart J. 2023 Apr;258:77-84. doi: 10.1016/j.ahj.2023.01.007. Epub 2023 Jan 13. PMID 36642225